CLINICAL TRIAL: NCT01257971
Title: Non-interventional Study to Assess Reaching of Cholesterol Target Values in Patients Treated With 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) Reductase Inhibitors in Croatia
Brief Title: Non-interventional Study (NIS) to Assess Reaching of Cholesterol Target Values in Patients Treated With HMG-CoA Reductase Inhibitors
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CHR-CRE-2010/1
Record Dates: First submitted 2010-12-06; First posted 2010-12-10 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Hypercholesterolaemia
Keywords: Cholesterol; HMG-CoA reductase inhibitor; cardiovascular risk; LDLl
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with hypercholesterolaemia

SUMMARY:
This is a multi-centre non-interventional study of patients who are treated with any HMGCoA reductase inhibitor available in Croatia (rosuvastatin, simvastatin, atorvastatin and fluvastatin) for at least 6 months. All HMG-CoA reductase inhibitors must be prescribed in accordance with SmPCs approved in Croatia. Data collection for each patient will take place at a single visit. The investigator will complete a Case Report Form with the patient's demographics, the presence of the factors for high cardiovascular risk, current treatment, cholesterol values as well as with further treatment decision.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been treated with one HMG-CoA reductase inhibitor for at least 6 months without changing the dose for the last 4 weeks at least.
* All patients must sign Informed consent form.

Exclusion Criteria:

* Patients who have not signed the Informed consent form.
* Patients with contraindication for the treatment with HMG-CoA reductase inhibitors as per SmPC approved in Croatia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by specialist
Sampling Method: Non-Probability Sample
Enrollment: 1868 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Number of patients reaching the LDL-C goals, according to the Fourth Joint European Task Force guideline | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated
Percentage of patients reaching the LDL-C goals, according to the Fourth Joint European Task Force guideline | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated

SECONDARY OUTCOMES:
Number of patients reaching the total cholesterol goals, according to the Fourth Joint European Task Force guideline. | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated
Number of patients with high cardiovascular risk reaching the LDL-C goals according to the Fourth Joint European Task Force guideline. | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated
Number of patients with high cardiovascular risk reaching the total cholesterol goals according to the Fourth Joint European Task Force guideline. | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated
Percentage of patients reaching the total cholesterol goals, according to the Fourth Joint European Task Force guideline. | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated
Percentage of patients with high cardiovascular risk reaching the LDL-C goals according to the Fourth Joint European Task Force guideline. | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated
Percentage of patients with high cardiovascular risk reaching the total cholesterol goals according to the Fourth Joint European Task Force guideline. | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated

CONTACTS AND LOCATIONS:
Overall Officials: Svjetlana Serdar, Study Chair — AstraZeneca; Karin Otter, Study Director — AstraZeneca
Locations (27):
- Croatia (27):
  - Research Site, Biograd na Moru
  - Research Site, Bjelovar
  - Research Site, Crikvenica
  - Research Site, Čakovec
  - Research Site, Dubrovnik
  - Research Site, Gospić
  - Research Site, Karlovac
  - Research Site, Koprivnica
  - Research Site, Krapina
  - Research Site, Krapinske Toplice
  - Research Site, Opatija
  - Research Site, Osijek
  - Research Site, Poreč
  - Research Site, Pula
  - Research Site, Rijeka
  - Research Site, Sisak
  - Research Site, Slavonski Brod
  - Research Site, Split
  - Research Site, Stubičke Toplice
  - Research Site, Umag
  - Research Site, Vinkovci
  - Research Site, Virovitica
  - Research Site, Virovitica- Slatina
  - Research Site, Vukovar
  - Research Site, Zadar
  - Research Site, Zageb
  - Research Site, Zagreb